## **Research Title:**

The Effect of Non-pharmacological (Exercise home-based method) intervention on psychological distress of patients undergoing hemodialysis at Al Suwaiq renal dialysis center.

NCT07083843

Date:

30/08/2024

## **Consent Form**

| Research title: The effect of Non-pharmacological intervention (exercises) on psychological distress of patient undergoing hemodialysis at ALSUWAIQ RENAL DIALYSIS CENTER. I, agree to participate in the research project, conducted by researcher, Amal AlSahi who has discussed the research project with me. | |
|---|---|
| I conse | nt to participate in the research project and the following has been explained to me: |
| > | the research may not be of direct benefit to me my participation is completely voluntary my right to withdraw from the study at any time without any implications to me the risks including any possible inconvenience, discomfort or harm as a consequence of my participation in the research project the steps that have been taken to minimize any possible risks what I am expected and required to do whom I should contact for any complaints with the research or the conduct of the research. I am able to request a copy of the research findings and reports Security and confidentiality of my personal information. Sion, I consent to: Publication of results from this study on the condition that my identify will not be revealed. |
| Name: | |
| Signatu | re: |
| Date: | |